CLINICAL TRIAL: NCT07120178
Title: Imaging and Evolution of Pigmented Tumors of the Anterior Ocular System in Children
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN222025/CHUSTE
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pigmented Tumours of the Anterior Ocular System in Children
Keywords: pigmented tumours of the anterior ocular system in children; CONJUNCTIVAL TUMORS CHILDREN
MeSH Terms: interventions — Slit Lamp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Children with pigmented tumors of the anterior ocular system
  Interventions: Other: slit lamp examination; Other: dermatoscopy examination x20 and x400; Other: confocal microscopy examination

INTERVENTIONS:
Other: slit lamp examination — data collected: tumor size, pigmentation, vascularization, cells
Other: dermatoscopy examination x20 and x400 — data collected: tumor size, pigmentation, vascularization, cells
Other: confocal microscopy examination — data collected: tumor size, pigmentation, vascularization, cells

SUMMARY:
The investigators were interested in pigmented tumours of the anterior segment of the eye in children because there is very little data on their evolution. The nevus is the most common conjunctival tumour.

The challenge is to be able to adapt the child's follow-up according to the imaging and avoid an invasive procedure such as surgical excision if the imaging does not find any suspicious cells despite a change in size or colour. This would also make it possible to answer parents' questions about the potential evolution of the tumour. Finally, it would enable the frequency of monitoring to be personalised according to the data analysed. The tests are all non-invasive and painless.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had a first dermato-ophthalmological consultation < 18 years old with pigmented tumors of the anterior ocular system

Exclusion Criteria:

* patient over 18 years old at first examination

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with pigmented tumors of the anterior ocular system
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The size and pigmentation of the tumor | Day 1
  Measurement of the size of the tumor with dermatoscopy x20 in mm and pigmentation with the slit lamp as well as dermatoscopy x20 and x400

SECONDARY OUTCOMES:
Describe the evolution according to age | Day 1
  Data collected from medical records
Describe the evolution according to sex | Day 1
  Data collected from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc PERROT, Md, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No